CLINICAL TRIAL: NCT06199115
Title: Prevention of Neuropathic Pain From Oxaliplatin by Photobiomodulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saint-Gregoire Private Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Neurosudoscan
Record Dates: First submitted 2023-12-21; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Cancer of the Gastrointestinal Tract
Keywords: Photobiomodulation; Pain; oxaliplatin; peripheral neuropathy; chemotherapy; SUDOSCAN
MeSH Terms: conditions — Gastrointestinal Neoplasms; Pain; Peripheral Nervous System Diseases | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients will not receive any intervention during their oxaliplatin chemotherapy cycles.
- Experimental (Experimental): Patients will receive three photobiomodulation sessions per week during their oxaliplatin chemotherapy cycles
  Interventions: Procedure: Photobiomodulation

INTERVENTIONS:
Procedure: Photobiomodulation — In oncology, photobiomodulation is used to help heal damaged tissues, improve immune response, reduce inflammation, and prevent or treat certain side effects of treatments such as chemotherapy. Photobiomodulation is also the subject of recent clinical studies to expand its indications (peripheral neuropathies induced by certain chemotherapies.
  Patients in the experimental group will receive 3 photobiomodulation sessions per week during their oxaliplatin treatments (6 months), for a total of 72 sessions. Exposition to laser light is 30 minutes for each session.
  Arms: Experimental

SUMMARY:
Peripheral neuropathy is one of the most common side effects of oxaliplatin (OXA)-based chemotherapy for patients treated for digestive cancers, disabling and dose-limiting. Several strategies have been studied for the treatment of oxaliplatin-related sensory neuropathy. Several pharmacological and non-pharmacological therapeutic strategies have been explored to relieve peripheral neuropathic pain. Non-pharmacological interventions have been shown to be potentially beneficial for patients suffering from chemotherapy-induced neurotoxicity. The objective of this prospective study is to evaluate the effectiveness of photobiomodulation on the reduction of neuropathic pain in patients who developed painful, cumulative peripheral neuropathy that appeared under the effect of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Recent diagnosis of digestive cancer
* 12 planned cycles of oxaliplatin
* Ability to understand and willingness to sign an informed consent form before starting any study procedures
* Patient benefiting from French health insurance

Exclusion Criteria:

* History of neuropathy before the start of the study,
* Symptomatic treatment of pain (or neuropathic pain),
* Patient with a psychotic disorder,
* Patient with diabetic neuropathy,
* Patient with metastatic cancer
* Patient with renal insufficiency,
* Adults under guardianship or curatorship,
* Vulnerable people

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Neuropathic Pain Synptom Inventory : pain | day 30, day 60, day 90, day 120, day 150, day 180, day 270
  Is is a score with 12 items. 10 items concern pain and are scale from 0 (no pain) to 10 (maximal pain).

SECONDARY OUTCOMES:
Health-relative quality of life of cancer patients participating to a clinical trial | day 0, day 60, day 120, day 180, day 270
  QLQ-C30 EORTC scale : 30 items scored from 1 (not at all) to 4 (very). Global health status, functional scales and symptom scales are reported.
Peripheral neuropathy : SUDOSCAN evaluation | day 0, day 30, day 60, day 90, day 120, day 150, day 180, day 270
  Evaluation of peripheral neuropathy by SUDOSCAN (detection and evaluation of small fiber neuropathies)
Peripheral neuropathy : electroneuromyogram evaluation | day 0, day 90, day 270
  Evaluation by electroneuromyogram : measurement of nerve conduction velocity
Evaluation of sensitive and motor symptoms | day 30, day 60, day 90, day 120, day 150, day 180, day 270
  TNSc score : 7 items to explore sensitive and motor symptoms, scored from 0 (no symptom) from 4 (very important symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Morgane Pihan, Principal Investigator — CHP Saint-Grégoire
Locations (1):
- CHP Saint-Grégoire, Saint-Grégoire, France

IPD SHARING:
Plan to Share IPD: No